CLINICAL TRIAL: NCT02094586
Title: Phase 3 Randomized, Double-blind, Placebo-Controlled 3-Lot Study in Healthy Volunteers to Assess Immunogenicity, & Acceptability of a Single-dose of Live Oral Cholera Vaccine, Vibrio Cholerae O1 Serotype Inaba Vaccine Strain CVD 103-HgR
Brief Title: A Phase 3 Lot to Lot Consistency Study of Live Oral Cholera Vaccine, PXVX0200 in Healthy Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bavarian Nordic (Industry)
Collaborators: Emergent BioSolutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PXVX-VC-200-004
Record Dates: First submitted 2014-03-20; First posted 2014-03-24 (Estimated); Results first posted 2021-07-15 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Cholera
MeSH Terms: conditions — Cholera

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- PXVX0200 Lot A (Experimental): PXVX0200 (Lot P700-1CA03) Single dose; liquid suspension after reconstitution with buffer; > 2x10^8 CFU in a liquid suspension
  Interventions: Biological: PXVX0200 Lot A
- PXVX0200 Lot B (Experimental): PXVX0200 (Lot P700-3CA03) Single dose; liquid suspension after reconstitution with buffer; > 2x10^8 CFU in a liquid suspension
  Interventions: Biological: PXVX0200 Lot B
- PXVX0200 Lot C (Experimental): PXVX0200 (Lot P700-6BA03) Single dose; liquid suspension after reconstitution with buffer; > 2x10^8 CFU in a liquid suspension
  Interventions: Biological: PXVX0200 Lot C
- Placebo (Placebo Comparator): Placebo physiological saline
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: PXVX0200 Lot A — Lot P700-1CA03
  Arms: PXVX0200 Lot A
Biological: PXVX0200 Lot B — Lot P700-3CA03
  Arms: PXVX0200 Lot B
Biological: PXVX0200 Lot C — Lot P700-6BA03
  Arms: PXVX0200 Lot C
Biological: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The primary goal of this Phase III study is to compare 3 lots for consistency of manufacture.

DETAILED DESCRIPTION:
The primary goal of this Phase III study is to compare three lots for consistency of manufacture.

ELIGIBILITY:
Inclusion Criteria:

* healthy men or women,
* age 18 to 45 years inclusive;
* normal medical history and physical examination
* Women must have a negative pregnancy test.

Exclusion Criteria:

* travel to a cholera endemic area in the previous 5 years;
* abnormal stool pattern or regular use of laxatives;
* Currently active unstable or undiagnosed medical conditions
* current or recent antibiotic use;
* pregnancy or nursing;
* Previously received a licensed or investigational cholera vaccine
* History of cholera or enterotoxigenic E. coli infection
* History of Guillain-Barré Syndrome
* Received or plans to receive any other licensed vaccines, except for seasonal influenza
* Recipient of bone marrow or solid organ transplant
* Malignancy (excluding non-melanotic skin cancers) or lymphoproliferative disorders diagnosed or treated during the past 5 years
* Use of systemic chemotherapy in the previous 5 years prior to the study
* any immunosuppressive medical condition

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3146 (Actual)
Dates: Start 2014-05; Primary Completion 2015-02 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James McCarty, MD, Study Director — Emergent Travel Health Inc.
Locations (25):
- United States (19):
  - Coastal Clinical Research, Mobile, Alabama
  - Clinical Reseach Consortium Arizona, Phoenix, Arizona
  - Avail Clinical Research, DeLand, Florida
  - Miami Research Associates, Miami, Florida
  - Palm Beach Research, West Palm Beach, Florida
  - Emory University, Atlanta, Georgia
  - Johnson County Clin-Trials, Lenexa, Kansas
  - Heartland Research Associates, Wichita, Kansas
  - Central Kentucky Research, Lexington, Kentucky
  - University of Kentucky, Lexington, Kentucky
  - Boston University, Boston, Massachusetts
  - Center for Pharmaceutical Research, Kansas City, Missouri
  - St. Louis University, St Louis, Missouri
  - Clinical Research Consortium Las Vegas, Las Vegas, Nevada
  - Rochester Clinical Research, Rochester, New York
  - Lion Research, Norman, Oklahoma
  - Coastal Carolina Research, Mt. Pleasant, South Carolina
  - Research Across America, Dallas, Texas
  - Jean Brown Research, Salt Lake City, Utah
- Australia (6):
  - QIMR Berghofer Medical Research Institiue, Herston, Queensland
  - AUS Trials Pty Ltd, Sherwood, Queensland
  - CMAX, Adelaide, South Australia
  - Emeritis Research, Malvern East, Victoria
  - Nucleus Network, Melbourne, Victoria
  - Linear Clinical Research, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] McCarty JM, Lock MD, Hunt KM, Simon JK, Gurwith M. Safety and immunogenicity of single-dose live oral cholera vaccine strain CVD 103-HgR in healthy adults age 18-45. Vaccine. 2018 Feb 1;36(6):833-840. doi: 10.1016/j.vaccine.2017.12.062. Epub 2018 Jan 6. PMID 29317118

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Following assignment to either receive PXVX0200 or placebo, subjects in the PXVX0200 arm were randomized to receive Lot A, B or C. Subjects in each of these Arms/Groups add up to the number of subjects in the PXVX0200 (Lot A, B and C) Arm/Group.
Groups:
- PXVX0200 Lot A; PXVX0200 Lot B; PXVX0200 Lot C: PXVX0200 Single dose; liquid suspension after reconstitution with buffer; 1x10^9 CFU in a liquid suspension
Period: Overall Study
Arm/Group | PXVX0200 Lot A | PXVX0200 Lot B | PXVX0200 Lot C | Placebo
Started | 927 | 933 | 935 | 351
Completed (Study Completion (Day 181) - Completion of study is based upon the Study Completion/Early Term eCRF) | 848 | 866 | 876 | 331
Not Completed | 79 | 67 | 59 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PXVX0200 Lot A | PXVX0200 Lot B | PXVX0200 Lot C | Placebo | Total
Number analyzed (Participants) | 927 | 933 | 935 | 351 | 3146
Age, Categorical [Count of Participants; unit: Participants]
  Between 18 and 45 years inclusive: <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 45 years inclusive: Between 18 and 65 years | 927 | 933 | 935 | 351 | 3146
  Between 18 and 45 years inclusive: >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.8 (7.78) | 29.9 (7.54) | 30.2 (7.72) | 29.5 (7.54) | 29.9 (7.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 510 | 503 | 514 | 155 | 1682
  Male | 417 | 430 | 421 | 196 | 1464
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 5 | 2 | 1 | 13
  Asian | 13 | 27 | 19 | 5 | 64
  Native Hawaiian or Other Pacific Islander | 3 | 2 | 3 | 1 | 9
  Black or African American | 222 | 238 | 231 | 115 | 806
  White | 649 | 626 | 655 | 218 | 2148
  More than one race | 20 | 20 | 14 | 7 | 61
  Unknown or Not Reported | 15 | 15 | 11 | 4 | 45
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 809 | 805 | 817 | 300 | 2731
  Australia | 118 | 128 | 118 | 51 | 415

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Ratio (GMR) at Day 11 for Vaccine Lots A and B
Description: The primary analysis consisted of three between-lot equivalence tests of serum vibriocidal antibody titer measured at Day 11. The GMT of each lot - µA, µB, and µC - was calculated by first log-transforming (base 10) the serum vibriocidal antibody titers, computing the means of the transformed data by lot, and then exponentiating the log-scale means to return to the original, untransformed scale. The resulting GMTs were combined to form three geometric mean ratios: µA/µB, µA/µC, and µB/µC.The ratios were required to be within +/- 50% of each other lot with 95% confidence, which implied that the limits of the 95% confidence interval on each pairwise GMR had to be within 0.67 - 1.5. Placebo GMT values were not included in the primary analysis.
Time Frame: Day 11
Population: The Immunogenicity Evaluable Population (IEP) comprises all randomized subjects who had evaluable vibriocidal antibody results from Day 11 and had no major protocol violations that affected immunogenicity.
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric Mean Titer
Groups:
- PXVX0200 Lot A; PXVX0200 Lot B: A single dose PXVX0200; liquid suspension after reconstitution with buffer; 1x10^9 CFU in a liquid suspension
Arm/Group | PXVX0200 Lot A | PXVX0200 Lot B
Number analyzed (Participants) | 892 | 887
Geometric Mean Titer | 9220 [8219 to 10343] | 10034 [8942 to 11260]
Statistical Analysis 1: Comparison: PXVX0200 Lot A; Lot A vs. Lot B; Test type: Equivalence — The GMT of each lot was required to be within ±50% of each other lot with 95% confidence. Specifically, the 95% CI around each pairwise ratio of GMTs was required to be within [0.67, 1.5]; Geometric Mean Ratio = 0.92, 95% CI 2-sided [0.78 to 1.08]

2. Secondary Outcome: SVA Seroconversion at Day 11
Description: Percentage of subjects who demonstrated a ≥4-fold rise over baseline in serum vibriocidal antibody (SVA) at Day 11
Time Frame: Day 11
Population: IEP - comprises all randomized subjects who had evaluable vibriocidal antibody results from Day 11 and had no major protocol violations that affected immunogenicity
Measure: Number (95% Confidence Interval); unit: % of participants
Arm/Group | PXVX0200 Lot A | PXVX0200 Lot B | PXVX0200 Lot C | Placebo
Number analyzed (Participants) | 892 | 887 | 909 | 334
% of participants | 94 [92 to 96] | 93 [91 to 94] | 94 [92 to 95] | 4 [2 to 7]

3. Secondary Outcome: SVA and Anti-CT IgG GMT at Day 1, 11, 29, 91 and 181
Description: GMTs of vibriocidal antibody and anti-CT IgG concentrations at Days 1, 11, 29, 91, and 181.
Time Frame: Day 1 - 181
Population: The subgroup examining long-term and specific functional immunogenicity was formed to examine specific behavior of Vaxchora based a smaller total sample size than the total study due to the complexity of the assays needed for the endpoints. As such, an analysis by lot would have rendered any examination severely underpowered and was not necessary due to the objective to examine Vaxchora vs placebo rather than the affect of lot on those endpoints.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Groups:
- PXVX0200 (Lot A, B and C): PXVX0200 Single dose; liquid suspension after reconstitution with buffer; 1x10^9 CFU in a liquid suspension
Arm/Group | PXVX0200 (Lot A, B and C) | Placebo
Number analyzed (Participants) | 26 | 6
Titer
  SVA GMT at Day 1 | 91 [52 to 162] | 143 [12 to 1728]
  SVA GMT at Day 11: number analyzed (Participants) | 22 | 4
  SVA GMT at Day 11 | 9922 [4306 to 22865] | 320 [6 to 16216]
  SVA GMT at Day 29 | 6170 [3798 to 10025] | 127 [10 to 1623]
  SVA GMT at Day 91 | 560 [322 to 975] | 127 [10 to 1623]
  SVA GMT at Day 181: number analyzed (Participants) | 26 | 5
  SVA GMT at Day 181 | 386 [211 to 703] | 53 [8 to 348]
  Anti-CT IgG GMT at Day 1 | 445 [405 to 489] | 951 [296 to 3057]
  Anti-CT IgG GMT at Day 11 | 1780 [901 to 3517] | 800 [319 to 2008]
  Anti-CT IgG GMT at Day 29 | 2007 [1075 to 3748] | 848 [316 to 2275]
  Anti-CT IgG GMT at Day 91 | 1276 [771 to 2111] | 599 [370 to 972]
  Anti-CT IgG GMT at Day 181: number analyzed (Participants) | 26 | 5
  Anti-CT IgG GMT at Day 181 | 1116 [687 to 1814] | 528 [329 to 846]

4. Secondary Outcome: SVA and Anti-CT IgG Seroconversion at Day 1, 11, 29, 91 & 181
Description: Proportion of subjects who demonstrated a ≥4-fold rise over baseline in vibriocidal antibody and anti-CT IgG concentration from baseline at Days 1, 11, 29, 91, and 181. Day 1 not reported as seroconversion on Day 1 not applicable.
Time Frame: Day 1 - 181
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: % of participants
Groups:
- PXVX0200: PXVX0200 Single dose; liquid suspension after reconstitution with buffer; 1x10^9 CFU in a liquid suspension
Arm/Group | PXVX0200 | Placebo
Number analyzed (Participants) | 26 | 6
% of participants
  SVA Seroconversion at Day 11: number analyzed (Participants) | 22 | 4
  SVA Seroconversion at Day 11 | 91 [71 to 99] | 0 [0 to 60]
  SVA Seroconversion at Day 29 | 96 [80 to 100] | 0 [0 to 46]
  SVA Seroconversion at Day 91 | 69 [48 to 86] | 0 [0 to 46]
  SVA Seroconversion at Day 181: number analyzed (Participants) | 26 | 5
  SVA Seroconversion at Day 181 | 50 [30 to 70] | 0 [0 to 52]
  Anti-CT IgG Seroconversion at Day 11 | 42 [23 to 63] | 0 [0 to 46]
  Anti-CT IgG Seroconversion at Day 29 | 46 [27 to 67] | 0 [0 to 46]
  Anti-CT IgG Seroconversion at Day 91 | 42 [23 to 63] | 0 [0 to 46]
  Anti-CT IgG Seroconversion at Day 181: number analyzed (Participants) | 26 | 5
  Anti-CT IgG Seroconversion at Day 181 | 35 [17 to 56] | 0 [0 to 52]

5. Secondary Outcome: Adverse Events
Description: Incidence and severity of signs and symptoms of reactogenicity such as diarrhea, fever & vomiting were collected from Day 1 - 8.
  Incidence and severity of unsolicited adverse events were collected till Day 29.
Time Frame: Day 1 - 29
Population: Safety population - the population of randomized subjects who received study treatment and was analyzed according to the treatment actually received.
Measure: Number; unit: % of participants
Groups:
- PXVX0200 (Lot A, B and C): PXVX0200 Single dose; liquid suspension after reconstitution with buffer; 1x10^9 CFU in a liquid suspension
  PXVX0200: comparing 3 lots of PXVX0200
Arm/Group | PXVX0200 Lot A | PXVX0200 Lot B | PXVX0200 Lot C | PXVX0200 (Lot A, B and C) | Placebo
Number analyzed (Participants) | 904 | 908 | 922 | 2734 | 350
% of participants
  % of Subjects with any Reactogenicity | 52.99 | 50.44 | 52.28 | 51.90 | 43.15
  % of Subjects with Diarrhea Symptoms | 4.31 | 3.96 | 3.36 | 3.88 | 1.17
  % of Subjects with Fever Symptoms | 0.77 | 0.77 | 0.33 | 0.62 | 1.17
  % of Subjects with Nausea/Vomiting | 18.03 | 18.94 | 18.00 | 18.32 | 15.16
  % of Subjects with Headache | 30.09 | 26.43 | 30.26 | 28.93 | 23.62

6. Primary Outcome: Geometric Mean Ratio (GMR) at Day 11 for Vaccine Lots B and C
Description: The primary analysis consisted of three between-lot equivalence tests of serum vibriocidal antibody titer measured at Day 11. The GMT of each lot - µA, µB, and µC - was calculated by first log-transforming (base 10) the serum vibriocidal antibody titers, computing the means of the transformed data by lot, and then exponentiating the log-scale means to return to the original, untransformed scale. The resulting GMTs were combined to form three geometric mean ratios: µA/µB, µA/µC, and µB/µC.The ratios were required to be within +/- 50% of each other lot with 95% confidence, which implied that the limits of the 95% confidence interval on each pairwise GMR had to be within 0.67 - 1.5.
Time Frame: Day 11
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric Mean Titer
Groups:
- PXVX0200 Lot C: A single dose PXVX0200; liquid suspension after reconstitution with buffer; 1x10^9 CFU in a liquid suspension
Arm/Group | PXVX0200 Lot B | PXVX0200 Lot C
Number analyzed (Participants) | 887 | 909
Geometric Mean Titer | 10034 [8942 to 11260] | 9827 [8770 to 11012]
Statistical Analysis 1: Comparison: PXVX0200 Lot B; Lot B vs Lot C; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Mean Ratio = 1.02, 95% CI 2-sided [0.87 to 1.20]

7. Primary Outcome: Geometric Mean Ratio (GMR) at Day 11 for Vaccine Lots A and C
Description: as for outcome 6
Time Frame: Day 11
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric Mean Titer
Groups:
- PXVX0200 Lot A; PXVX0200 Lot C: A of single dose PXVX0200; liquid suspension after reconstitution with buffer; 1x10^9 CFU in a liquid suspension
Arm/Group | PXVX0200 Lot A | PXVX0200 Lot C
Number analyzed (Participants) | 892 | 909
Geometric Mean Titer | 9220 [8219 to 10343] | 9827 [8770 to 11012]
Statistical Analysis 1: Comparison: PXVX0200 Lot A; Lot A vs. Lot C; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Geometric Mean Ratio = 0.94, 95% CI 2-sided [0.80 to 1.10]

ADVERSE EVENTS:
Time Frame: Unsolicited AEs, serious adverse events (SAEs), medically attended events, and new onset of chronic medical conditions were assessed for 180 days post-vaccination.
Description: Totals presented are the number of subjects with at least one AE. Analysis of all cause mortality, SAEs and other serious events were performed for the safety population (N=2789) and not the randomized population. Only the SAEs were analyzed per lot while the analysis for the AEs was not completed for subjects that received each lot. This covers the entire safety of Vaxchora to provide the overall profile. The larger sample size afforded better estimates of risk for the observed events.
Groups:
- All PXVX0200 Lots: All PXVX0200 Lots
Arm/Group | PXVX0200 Lot A | PXVX0200 Lot B | PXVX0200 Lot C | All PXVX0200 Lots | Placebo
All-Cause Mortality (participants affected / at risk) | 1/926 | 0/928 | 0/935 | 1/2789 | 0/350
Serious Adverse Events (participants affected / at risk) | 7/926 | 9/928 | 4/935 | 20/2789 | 3/350
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 290/2789 | 33/350
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PXVX0200 Lot A (N=926) | PXVX0200 Lot B (N=928) | PXVX0200 Lot C (N=935) | All PXVX0200 Lots (N=2789) | Placebo (N=350)
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 2 | 0 | 2 | 0
Kidney Infection (Infections and infestations) | 0 | 1 | 0 | 1 | 1
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Ankle Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 | 0
Jaw Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
Patella Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
Stress Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0
Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0 | 1 | 0
Completed Suicide (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PXVX0200 Lot A (N=0) | PXVX0200 Lot B (N=0) | PXVX0200 Lot C (N=0) | All PXVX0200 Lots (N=2789) | Placebo (N=350)
Headache (Nervous system disorders) | NA | NA | NA | 75 | 11
Fatigue (General disorders) | NA | NA | NA | 59 | 8
Upper Respiratory Tract Infection (Infections and infestations) | NA | NA | NA | 57 | 5
Back Pain (Musculoskeletal and connective tissue disorders) | NA | NA | NA | 38 | 3
Flatulence (Gastrointestinal disorders) | NA | NA | NA | 32 | 4
Abdominal Pain (Gastrointestinal disorders) | NA | NA | NA | 29 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days